CLINICAL TRIAL: NCT01977560
Title: Diet and Exercise Intervention in Type 2 Diabetes
Acronym: LID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Dairy Council (Other); American Egg Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201302095
Record Dates: First submitted 2013-10-14; First posted 2013-11-06 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Exercise; Weight loss
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Weight Loss | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Other): Participants randomized to this arm will receive dietary and physical activity instructions as recommended by the American Diabetes Association (ADA) guidelines.
  Interventions: Behavioral: Standard Care
- Intensive Lifestyle intervention (Experimental): Participants randomized to this arm will be participate in weekly dietary and behavioral education session in addition to four 60-min supervised exercise training sessions per week for 8 months. All dietary and- behavioral education and exercise training sessions will be conducted at the worksite.
  Interventions: Behavioral: Intensive Lifestyle Intervention

INTERVENTIONS:
Behavioral: Intensive Lifestyle Intervention — Participants will be instructed to consume ~500 kcal/day less than their calculated estimated total daily energy requirements. The supervised exercise program will include both endurance and resistance exercise training sessions. The doses of diabetes medications will be adjusted by study physicians every 1-2 weeks, as needed to avoid hypoglycemia.
  Arms: Intensive Lifestyle intervention
Behavioral: Standard Care — After receiving dietary and physical activity instructions as recommended by the American Diabetes Association (ADA) guidelines participants will meet approximately every month for about 7 months with a study team member to record body weight, review diet and physical activity behaviors, and document medication use. Participants will continue their routine medical management, including regular clinic visits with their personal physician and/or diabetes educator during their participation in this study. Any changes medications will made by the participants' personal physician(s).
  Arms: Standard Care

SUMMARY:
The purpose of this study is to determine the effect of a worksite-based intensive lifestyle therapy intervention (weight loss with exercise training) on blood sugar control in people with obesity and type 2 diabetics.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a randomized, controlled trial in people with obesity and type 2 diabetes to determine the therapeutic effects of intensive lifestyle therapy conducted at the worksite compared to standard care on: i) the major factors involved in the pathogenesis of type 2 diabetes (insulin sensitivity, β-cell function and the metabolic response to glucose ingestion), ii) body composition; iii) physical function (cardiorespiratory fitness and muscle strength); iv) and the potential cellular mechanisms that can affect insulin action in muscle and adipose tissue (fat).

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-68 yrs old
2. BMI 27.0-50.0 kg/m²
3. Diagnosis of type 2 diabetes based on HbA1C>6.5% or results of an oral glucose tolerance test or current use of anti-diabetic medications
4. HbA1C ≤9.5 %.
5. Work at Washington University in St. Louis, Barnes Jewish Hospital, St. Louis Children's Hospital, Shriners, St. Louis College of Pharmacy, Central Institute for the Deaf, Rehabilitation Institute of St. Louis, and/or any institutions affiliated with these.

Exclusion Criteria:

1. Any change in diabetes medication in previous 3 months
2. Treated with >0.5 units of insulin/kg body weight per day
3. Unstable weight (>2% change during the last 2 months before entering the study)
4. History or evidence of serious pulmonary or cardiovascular disease, including acute coronary syndrome, heart failure requiring medications, or New York Heart Association class III heart failure (patients with marked limitation of activity and who are comfortable only at rest) or IV heart failure (patients who should be at complete rest, confined to bed or chair and who have discomfort with any physical activity).
5. Evidence of serious cardiac abnormalities during exercise stress testing that increase cardiac risk of initiating an exercise program.
6. Creatinine >1.5 mg/dL
7. Microalbuminuria; spot urine albumin:creatinine ratio >50 (50 μg albumin/mg creatinine)
8. Coagulation disorders
9. Anemia (Hemoglobin <10.0 g/dL)
10. Liver enzymes (ALT and AST) ≥3 times the upper limit of normal
11. Uncontrolled proliferative diabetic retinopathy
12. Severe peripheral neuropathy diagnosed by monofilament testing
13. Severe organ dysfunction
14. Pregnant or breastfeeding
15. Participating in regular exercise (>1 h of structured exercise/week)
16. Joint replacement within the last year
17. Smokes tobacco
18. Severe lactose intolerance
19. Take any medication that might interfere with interpretation of the metabolic studies
20. Unable or unwilling to follow the study protocol or for any reason the research team believes the volunteer is not an appropriate candidate for this study, including non-compliance with screening appointments or previous medical visits.

Ages: 25 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle insulin sensitivity | 7-8 months
  Skeletal muscle insulin sensitivity will be calculated as the glucose disposal rate per kg fat-free mass divided by plasma insulin during a hyperinsulinemic-euglycemic clamp procedure.

SECONDARY OUTCOMES:
Liver insulin sensitivity | 7-8 months
  Liver insulin sensitivity will be assessed by using the hepatic insulin sensitivity index.
Adipose tissue insulin sensitivity | 7-8 months
  Adipose tissue insulin sensitivity will be assessed by using the adipose tissue insulin sensitivity index.
β-cell function | 7-8 months
  β-cell function will be assessed from a modified oral glucose tolerance test
Insulin clearance | 7-8 months
  Insulin clearance will be assessed from a modified oral glucose tolerance test
Diabetes remission | 7-8 months
  Remission of type 2 diabetes will be defined as HbA1c <6.0% without the use of diabetes medications use of diabetes medications.
Cardiorespiratory fitness | 7-8 months
  Peak oxygen consumption will be assessed using indirect calorimetry during a graded exercise test to volitional exhaustion.
Muscle strength | 7-8 months
  Muscle strength will be assessed as the total maximal weight lifted during the 1 repetition maximum tests for leg press, knee flexion, seated row, and chest press exercises.
Whole-body fat mass | 7-8 months
  Total body fat mass will be assessed by dual-energy X-ray absorptiometry.
Whole-body fat-free mass | 7-8 months
  Fat-free mass will be assessed by dual-energy X-ray absorptiometry.
Appendicular lean mass | 7-8 months
  Appendicular lean mass will be assessed by dual-energy X-ray absorptiometry.
Intra-abdominal adipose tissue volume | 7-8 months
  Intra-abdominal adipose tissue volume will be determined by using magnetic resonance imaging.
Intrahepatic triglyceride content | 7-8 months
  Intrahepatic triglyceride content will be determined by using magnetic resonance spectroscopy.
Plasma adipokine concentrations | 7-8 months
  Plasma adiponectin and PAI-1 concentrations will be measured in the Washington University Clinical Core Laboratory.
Transcriptome in muscle and adipose tissue | 7-8 months
  The transcriptome (all RNA that are responsible for making proteins from DNA templates) will be evaluated by using RNA sequencing techniques.
Skeletal muscle mitochondrial metabolites | 7-8 months
  The content of muscle mitochondrial-related metabolites will be determined by liquid chromatography mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Yoshino M, Yoshino J, Smith GI, Stein RI, Bittel AJ, Bittel DC, Reeds DN, Sinacore DR, Cade WT, Patterson BW, Cho K, Patti GJ, Mittendorfer B, Klein S. Worksite-based intensive lifestyle therapy has profound cardiometabolic benefits in people with obesity and type 2 diabetes. Cell Metab. 2022 Oct 4;34(10):1431-1441.e5. doi: 10.1016/j.cmet.2022.08.012. Epub 2022 Sep 8. PMID 36084645
- [Derived] Mittendorfer B, Patterson BW, Smith GI, Yoshino M, Klein S. beta Cell function and plasma insulin clearance in people with obesity and different glycemic status. J Clin Invest. 2022 Feb 1;132(3):e154068. doi: 10.1172/JCI154068. PMID 34905513